CLINICAL TRIAL: NCT05182723
Title: Evaluation of the Effectiveness of Extracorporeal Methods for Removing Mediators of Systemic Inflammation in Patient With Multiple Organ Dysfunction Syndrome After Heart and Aortic Surgery
Brief Title: Evaluation of the Effectiveness of Extracorporeal Methods for Removing Mediators of Systemic Inflammation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Petrovsky National Research Centre of Surgery (Other)
Responsible Party: Principal Investigator, Aleksandr Eremenko, Clinical Professor, Petrovsky National Research Centre of Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20211028-18
Record Dates: First submitted 2021-12-01; First posted 2022-01-10 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Renal Failure Acute; Multiple Organ Failure; Cardiovascular Diseases
Keywords: mediators of systemic inflammation; extracorporeal methods; interleukins
MeSH Terms: conditions — Acute Kidney Injury; Multiple Organ Failure; Cardiovascular Diseases | interventions — Renal Replacement Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oXiris (Active Comparator): Monotoring of extracorporeal Method for Removing Mediators of Systemic Inflammation of oXiris will be performed for 24 hours
  Interventions: Procedure: renal replacement therapy
- oXiris in combination with Jafron HA330 (Experimental): Extracorporeal Method for Removing Mediators of Systemic Inflammation oXiris in combination with Jafron HA330 will be performed for 4 hours.
  If SOFA is more or equally 4 , CRP is more than 100 ng/ml;, the IL6 value is increased by 5 or more times after 12 hours of procedure Jafron HA330 will be reconnected and performed for 4 hours.
  Monitoring of whole procedure will be performed for 24 hours.
  Interventions: Procedure: renal replacement therapy

INTERVENTIONS:
Procedure: renal replacement therapy — Extracorporeal Methods for Removing Mediators of Systemic Inflammation

SUMMARY:
The purpose of this study is to assess the effectiveness and the safety of extracorporeal methods for removing mediators of systemic inflammation in patients with multiple organ dysfunction syndrome after heart and aorta surgery.

DETAILED DESCRIPTION:
After being informed about the study and potential risk, all patients with multiple organ dysfunction syndrome after heart and aorta surgery with indications for extracorporeal removal of inflammatory mediators, giving written informed consent will be included in the study.

Patients will be randomized 1:1 ratio to 1. hemoperfusion cartridge for cytokine sorption in combination with an oXiris membrane and 2. oXiris membrane.

ELIGIBILITY:
Inclusion Criteria:

* multiple organ dysfunction;
* SOFA equal to or more than 4;
* CRP equal to or more than 100 ng / ml;
* increase of IL6 by 5 times or more

Exclusion Criteria:

* the impossibility to use heparin ( bleeding; heparin-induced thrombocytopenia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-25 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
CRP | 12 hours from the beginning of the study
  сhange of CRP after 12 hours from baseline value
CRP | 24 hours from the beginning of the study
  сhange of CRP after 24 hours from baseline value
CRP | 24 hours from the beginning of the study
  comparison of CRP after 12 hours with CRP after 24 hours
IL6 | 12 hours from the beginning of the study
  сhange of IL6 after 12 hours from baseline value
IL6 | 24 hours from the beginning of the study
  сhange of IL6 after 24 hours from baseline value
IL6 | 24 hours from the beginning of the study
  comparison of IL6 after 12 hours with IL6 after 24 hours
SOFA | 12 hours from the beginning of the study
  change of SOFA values after 12 hours from baseline value
SOFA | 24 hours from the beginning of the study
  change of SOFA values after 24 hours from baseline value
SOFA | 24 hours from the beginning of the study
  comparison of the SOFA value after 12 hours with the SOFA value after 24 hours

SECONDARY OUTCOMES:
extracorporeal therapy | hospitalisation period, an average of 1 month
  duration
time spent in intensive care unit | hospitalisation period, an average of 1 month
  duration
inpatient stay time | through study completion, an average of 2 months
  duration
renal function of RIFLE | through study completion, an average of 2 months
  percentage decrease from initial level
lethality | through study completion, an average of 2 months
  ratio of the number of deaths to the total number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandr Eremenko, MD, Study Director — Petrovsky National Research Centre of Surgery; Tatiana Marchenko, Principal Investigator — Petrovsky National Research Centre of Surgery
Locations (1):
- Petrovsky Nacional research Centre of Surgery, Moscow, Russia